CLINICAL TRIAL: NCT07351474
Title: Effect of Remimazolam on Postoperative Delirium in Elderly Patients Undergoing Laparoscopic Radical Gastrectomy: A Prospective Randomized Controlled Trial
Brief Title: Remimazolam for Reducing Postoperative Delirium in Elderly Patients Undergoing Laparoscopic Gastrectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xiongxiong Pan, Associate Chief Physician, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-SR-1025
Record Dates: First submitted 2025-12-14; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer; Postoperative Delirium
Keywords: Remimazolam; Propofol; Elderly Patients; Laparoscopic Gastrectomy; Anesthesia; Postoperative Delirium
MeSH Terms: conditions — Stomach Neoplasms; Emergence Delirium | interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam Group (Experimental): Participants in this group will receive remimazolam for anesthesia induction and maintenance during laparoscopic radical gastrectomy.
  Interventions: Drug: Remimazolam
- Propofol Group (Active Comparator): Participants in this group will receive propofol for anesthesia induction and maintenance during laparoscopic radical gastrectomy.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — Remimazolam will be used as the primary anesthetic agent for induction and maintenance. Dosage will be adjusted to maintain BIS between 40 and 60.
  Arms: Remimazolam Group
Drug: Propofol — Propofol will be used as the primary anesthetic agent for induction and maintenance. Dosage will be adjusted to maintain BIS between 40 and 60.
  Arms: Propofol Group

SUMMARY:
This prospective, randomized controlled clinical trial aims to evaluate whether remimazolam can reduce the incidence of postoperative delirium (POD) in elderly patients undergoing laparoscopic radical gastrectomy for gastric cancer. A total of 170 patients aged 65 years or older will be enrolled and randomized in a 1:1 ratio to receive either remimazolam or a propofol-midazolam regimen for anesthesia induction and maintenance. Standard perioperative monitoring, BIS-guided anesthesia depth control, and postoperative pain management will be applied in both groups. The primary outcome is the incidence of postoperative delirium within 5 days after surgery, assessed twice daily using the 3D-CAM. Secondary outcomes include emergence agitation, extubation time, postoperative pain scores, cognitive function at discharge, intraoperative hemodynamic stability, unplanned ICU admission, postoperative complications, and length of ICU stay. This study aims to determine whether remimazolam provides a safer and more effective anesthetic option for improving postoperative neurological outcomes and recovery in elderly patients undergoing laparoscopic radical gastrectomy.

DETAILED DESCRIPTION:
This prospective, randomized, controlled clinical trial is designed to investigate the efficacy and safety of remimazolam in reducing postoperative delirium (POD) among elderly patients undergoing laparoscopic radical gastrectomy. Postoperative delirium is a common and serious complication in older surgical patients and is associated with prolonged recovery, cognitive decline, increased morbidity, higher healthcare costs, and long-term mortality. Despite advances in perioperative care, effective strategies for reducing POD in elderly patients undergoing major abdominal surgery remain limited. Remimazolam, a novel ultra-short-acting benzodiazepine, offers rapid metabolism, hemodynamic stability, and reliable reversibility, making it a potentially advantageous anesthetic agent for this high-risk patient population.

A total of 170 eligible patients aged 65 years or older will be enrolled at The First Affiliated Hospital of Nanjing Medical University. Participants will be randomized in a 1:1 ratio to receive either remimazolam (R group) or a propofol-midazolam regimen (P group) during anesthesia induction and maintenance. Randomization will be performed using a computer-generated sequence and sealed opaque envelopes. Anesthesia depth will be monitored by BIS, and drug dosages will be dynamically adjusted to maintain BIS between 40 and 60 while keeping hemodynamic parameters within 20% of baseline values. Standardized perioperative management will be applied to all participants, including opioid analgesia, muscle relaxation, controlled ventilation, vasoactive medication titration, and postoperative PCIA.

Postoperative delirium will be assessed twice daily from postoperative day 1 to day 5 using the 3D-CAM diagnostic criteria by trained evaluators blinded to group allocation. Delirium assessments will also be conducted on the day of surgery at least two hours after emergence. Additional postoperative evaluations will include pain scores (NRS), emergence agitation, MMSE cognitive assessments, extubation time, PACU duration, length of hospitalization, and adverse events such as intraoperative awareness, hypotension, postoperative nausea and vomiting, or unplanned ICU admission.

Intraoperative data-including anesthesia duration, surgical duration, anesthetic drug dosages, opioid consumption, vasoactive medication use (converted to norepinephrine-equivalent doses), fluid balance, and estimated blood loss-will be recorded. Preoperative data collection includes demographics, comorbidities, Charlson Comorbidity Index, medication history, laboratory findings, and sleep quality. Data collection will continue until postoperative day 5 or hospital discharge, whichever occurs first.

The primary outcome of this trial is the incidence of postoperative delirium within five days after surgery. Secondary outcomes include the severity and subtype of delirium, emergence agitation, cognitive function at discharge, postoperative pain scores, extubation time, postoperative complications, PACU stay, ICU stay, and length of hospitalization. Statistical analyses will be conducted by investigators blinded to group allocation using standard tests for normality, t-tests or Mann-Whitney U tests for continuous variables, and Chi-square or Fisher exact tests for categorical variables. A two-sided P value <0.05 will be considered statistically significant.

This study is expected to provide evidence regarding whether remimazolam offers superior neurocognitive outcomes, improved hemodynamic stability, and fewer postoperative complications compared with propofol-based anesthesia in elderly patients undergoing laparoscopic radical gastrectomy. The findings may support the development of safer anesthesia strategies and enhanced recovery protocols for elderly surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years.
* Body mass index (BMI) between 18 and 28 kg/m².
* ASA physical status I-III.
* Scheduled for elective laparoscopic radical gastrectomy under general anesthesia at Jiangsu Province Hospital.
* Able and willing to sign informed consent.

Exclusion Criteria:

* Severe respiratory, cardiovascular, renal, or hepatic dysfunction.
* Stroke within the past 6 months or other central nervous system diseases.
* History of schizophrenia, epilepsy, Parkinson's disease, myasthenia gravis, or other psychiatric disorders.
* History of alcohol abuse or psychoactive substance dependence.
* Severe visual, hearing, or language impairment preventing communication.
* Allergy or contraindication to propofol or benzodiazepines.
* Preoperative cognitive impairment assessed by MMSE (≤24 for ≥middle-school education; ≤20 for primary school; ≤17 for no formal education).
* Participation in another drug clinical trial within 1 month before surgery.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of Postoperative Delirium | From postoperative Day 1 to Day 3
  Postoperative delirium will be assessed using the 3D-CAM diagnostic tool by trained evaluators blinded to group assignment. Delirium will be identified based on the presence of acute onset/fluctuation, inattention, altered consciousness, or disorganized thinking, following the standard 3D-CAM algorithm.

SECONDARY OUTCOMES:
Emergence Agitation | Immediately after extubation until PACU discharge
  Emergence agitation will be assessed in the PACU using the RASS or agitation scale by blinded evaluators.
Time to extubation | At the end of surgery
  Time from discontinuation of anesthetic agents to successful tracheal extubation.
Postoperative Pain Score | At PACU discharge; postoperative day 1,day 2,and day 3.
  Pain itensity will be evaluated using the Numerical Rating Scale(NRS,0-10)
Post-induction Hypotension | From completion of anesthetic induction to 10 minutes after induction.
  Post-induction hypotension will be defined as a decrease in mean arterial pressure (MAP) to <65 mmHg or a reduction of ≥30% from baseline within the first 10 minutes after anesthetic induction.
Incidence of Postoperative Nausea and Vomiting | From surgery until 48 hours postoperatively
  Postoperative nausea and vomiting assessed as the presence or absence based on patient reports and medical records during the postoperative period.
Length of Hospital Stay(days) | From the day of surgery (Day 0) to the date of hospital discharge (expected within 7-14 days postoperatively)
  Length of hospital stay is defined as the number of calendar days from the date of surgery (Day 0) until the date of hospital discharge , as recorded in the electronic medical record system

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751